CLINICAL TRIAL: NCT01672606
Title: Effect of Partial Neuromuscular Blockade by Rocuronium on the Acute Hypoxic Ventilatory Response in Patients With Obstructive Sleep Apnea-before and After Three Month CPAP Treatment. A Non-randomized, Non-blinded Study.
Brief Title: Effect of Rocuronium on the Acute Hypoxic Ventilatory Response in Patients With Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malin Jonsson Fagerlund (Other)
Responsible Party: Sponsor-Investigator, Malin Jonsson Fagerlund, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSA ROC
Record Dates: First submitted 2012-06-01; First posted 2012-08-27 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: OSA; Rocuronium; Neuromuscular Blockade; Hypoxic Ventilatory Response; CPAP
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rocuronium (Experimental): Intravenous infusion of rocuronium with the goal of TOF 0.70 and >0.90
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — Partial neuromuscular blockade with rocuronium with a TOF 0.70
  Other Names: CPAP

SUMMARY:
This study describe the effect of partial neuromuscular blockade of rocuronium on the acute hypoxic ventilatory response in patients with OSA before and after 3 month of CPAP treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male with diagnosed moderate OSA (AHI 15-30), untreated, but planned for CPAP treatment. Healthy except for OSA and well controlled tablet treated hypertension where the treatment has not been changed during the last 3 month. None smokers. 18-70 years old. BMI <35.

Exclusion Criteria:

* If they don´t fit the inclusion criteria

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Hypoxic ventilatory response | At baseline, with CPAP, at TOF 0.70 and at TOF >0.90. At diagnosis and after 3 month of CPAP treatment at home

SECONDARY OUTCOMES:
Hypercarbic ventilatory response | At baseline, with CPAP, at TOF 0.70 and at TOF >0.90. At diagnosis and after 3 month of CPAP treatment at home
Hypoxic ventilatory response | At diagnosis and after 3 month of CPAP treatment at home
Hypoxic ventilatory response during acute CPAP treatment | At diagnosis and after 3 month of CPAP treatment
Hypercarbic ventilatory response | At diagnosis and after 3 month of CPAP treatment at home
Hypercarbic ventilatory response during acute CPAP treatment | At diagnosis and after 3 month CPAP treatment at home
Upper airway obstruction | At TOF 0.70 and TOF >0.90. At diagnosis and after 3 month CPAP treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Malin Jonsson Fagerlund, MD, PhD, Principal Investigator — Karolinska University Hospital and Karolinska Institutet
Locations (1):
- Department of Anesthesiology, Surgical Sciences and Intensive Care Medicine, Karolinska University Hospital, Stockholm, Sweden